CLINICAL TRIAL: NCT05263167
Title: Reducing Edema After intraCerebral Hemorrhage
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 100999
Record Dates: First submitted 2022-01-09; First posted 2022-03-02 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Edema Brain
Keywords: edema; intracerebral hemorrhage; sodium aescinate
MeSH Terms: conditions — Brain Edema; Edema; Cerebral Hemorrhage | interventions — sodium aescinate; Injections; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sodium aescinate group (Experimental): Trial treatment is administered as sodium Aescinate 10mg in 250ml sodium chloride 0.9% infusion bag intravenously once daily for 10 days.
  Interventions: Drug: Sodium Aescinate
- placebo group (Placebo Comparator): Trial treatment is administered as 250ml sodium chloride 0.9% infusion bag intravenously once daily for 10 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sodium Aescinate — sodium Aescinate 10mg in 250ml sodium chloride 0.9% infusion bag intravenously once daily for 10 days.
  Other Names: Sodium Aescinate for Injection
  Arms: sodium aescinate group
Drug: Placebo — 250ml sodium chloride 0.9% infusion bag intravenously once daily for 10 days.
  Other Names: 0.9% sodium chloride injection
  Arms: placebo group

SUMMARY:
The REACH trial is a prospective multicenter double-blind randomized placebo-controlled trial with blinded end-point adjudication. Participants are randomized (1:1) to receive either sodium aescinate or matching placebo (0.9% saline). The primary outcome is the absolute volume of PHE evaluated based on brain CT image on day 14 after ICH.

DETAILED DESCRIPTION:
The REACH trial is a prospective multicenter double-blind randomized placebo-controlled trial with blinded end-point adjudication. Participants are randomized (1:1) to receive either sodium aescinate or matching placebo (0.9% saline). The primary outcome is the absolute volume of PHE evaluated based on brain CT image on day 14 after ICH. Functional outcome is assessed face to face at 3-month after onset. Meanwhile, central telephone follow-up determines functional outcomes at 3-month after onset. Brain imaging (CT) is performed as part of routine care prior to enrolment. A research CT scan is performed after 24h of symptom onset to assess hematoma expansion; a second research CT scan is performed at 72 hours after onset to assess brain swelling and dynamic change of PHE. The study was approved by the ethics committee of the Beijing Tiantan hospital. The study is conducted according to GCP guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged between 18-80 years old;
2. Spontaneous ICH confirmed by cranial CT;
3. Time from onset to randomization within 24 hours;
4. Superatentorial ICH;
5. Hematoma volume between 10-30 ml (calculated using ABC/2 method);
6. Glasgow coma scale (GCS) > 9 on admission;
7. informed and consent.

Exclusion Criteria:

1. Suspected secondary cause of ICH (e.g. aneurysm, vascular malformation, neoplasia, cerebral venous thrombosis, hemorrhagic transformation of recent ischemic stroke, thrombolysis or endovascular treatment, anticoagulation, et al);
2. ICH secondary to trauma；
3. Primary intraventricular hemorrhage (IVH);
4. Signs of herniation, such as progressive decline in consciousness, decreased or disappearance of pupillary light reflection, bilateral pyramidal tract signs, etc;
5. Other serious, advanced or terminal illness such that life expectancy is less than one year (e.g. advanced metastatic cancer);
6. Severe cardiac insufficiency (NYHA class III or IV);
7. High-risk arrhythmia, such as sick sinus syndrome, second or third degree atrioventricular block, bradycardia-related syncope without a pacemaker, etc;
8. Severe liver insufficiency; severe liver insufficiency is defined as ALT > 2 times the upper limit of normal or AST greater than 2 times the upper limit of normal;
9. Severe renal insufficiency: Severe renal insufficiency is defined as creatinine greater than 1.5 times the upper limit of normal;
10. History of severe asthma or chronic obstructive pulmonary disease (COPD);
11. History of coagulopathy or systemic bleeding;
12. A thrombocyte count below <100 x 10^9/L or leukocytosis < 2 x 10^9/L on admission;
13. Patients who plan to undergo surgical intervention before the first administration, including but not limited to hematoma removal (including minimally invasive and conventional surgery), decompressive craniectomy, hematoma aspiration, and ventricular puncture external drainage;
14. Patients with preexisting disability of a modified Rankin Scale (mRS) score greater than 2 prior to ICH;
15. Unable to understand the research procedures and/or complete follow-up due to mental illness, cognitive impairment, affective disorder, etc;
16. Women of childbearing potential, pregnant, or breastfeeding at randomization;
17. Contraindication to sodium aescinate；
18. Participate in other clinical studies within 3 months or are participating in other clinical studies.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-03-15 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Absolute edema volume on day 14 after ICH | on day 14 after ICH
  Absolute edema volume is based on brain CT image

SECONDARY OUTCOMES:
Relative edema volume on day 14 after ICH | on day 14 after ICH
  Relative edema volume is based on edema volume divided by hematoma volume
Absolute edema volume and relative edema volume on 24 ±12 hour and 72±12 hour after ICH symptom onset | on 24±12 hour and 72±12 hour after ICH symptom onset
  absolute edema volume is based on brain CT image；relative edema volume is based on edema volume divided by hematoma volume
Cytotoxic edema on 72 ±12 hour after ICH symptom onset | on 72 ±12 hour after ICH symptom onset
  Cytotoxic edema is based on brain MRI image
Dynamic changes of serum IL-x levels(ng/ml) within 14 days of symptom onset | within 14 days of symptom onset
  The purpose is to evaluate dynamic changes of serum inflammatory factor levels within 14 days of symptom onset
Dynamic changes of serum NF-kB levels(ug/ml) within 14 days of symptom onset | within 14 days of symptom onset
  The purpose is to evaluate dynamic changes of serum inflammatory factor levels within 14 days of symptom onset
Dynamic changes of serum TNF levels(ng/ml) within 14 days of symptom onset | within 14 days of symptom onset
  The purpose is to evaluate dynamic changes of serum inflammatory factor levels within 14 days of symptom onset
Dynamic changes of serum MMPs levels(ug/ml) within 14 days of symptom onset | within 14 days of symptom onset
  The purpose is to evaluate dynamic changes of serum inflammatory factor levels within 14 days of symptom onset
Dynamic changes of serum VEGF levels(pg/ml) within 14 days of symptom onset | within 14 days of symptom onset
  The purpose is to evaluate dynamic changes of serum inflammatory factor levels within 14 days of symptom onset
Dynamic changes of serum EPO levels(ng/ml) within 14 days of symptom onset | within 14 days of symptom onset
  The purpose is to evaluate dynamic changes of serum inflammatory factor levels within 14 days of symptom onset
Dynamic changes of serum angiopoietin-1 levels(pg/ml) within 14 days of symptom onset | within 14 days of symptom onset
  The purpose is to evaluate dynamic changes of serum inflammatory factor levels within 14 days of symptom onset
Change of neurological dysfunction within 14 days of symptom onset | within 14 days of symptom onset
  Change of neurological dysfunction within 14 days of symptom onset is based on National institute of health stroke scale(NIHSS）14d-NIHSS enrollment.（The minimum and maximum values of NIHSS is 0 and 42,respectively, higher scores mean a worse outcome.）
Cognition（MMSE) at 14 days of symptom onset | at 14 days of symptom onset
  Cognition is based on Mini-mental State Examination（MMSE）. （The minimum and maximum values of MMSE is 0 and 30,respectively, higher scores mean a better outcome. ）
Cognition（MoCA) at 14 days of symptom onset | at 14 days of symptom onset
  Cognition is based on Montreal Cognitive Assessment（MoCA）. （The minimum and maximum values of MoCA is 0 and 30,respectively, higher scores mean a better outcome.）
Dependency at 90±7 days after onset | at 90±7 days after onset
  Dependency at 90±7 days after onset Dependency is based on Modified Rankin Scale（mRS ）.
  （The minimum and maximum values of mRS is 0 and 5,respectively, higher scores mean a worse outcome.）
Quality of life at 90±7 days after onset | at 90±7 days after onset
  Quality of Life is based on five-level version of EuroQol Five Dimensions Questionnaire（EQ-5D-5L）.
  （The scale mainly contains 5 dimensions, including mobility, self-care ability, ability to perform daily activities, pain or discomfort, and anxiety or depression. Each dimension is divided into 5 levels: no difficulty, mild difficulty, moderate difficulty, severe difficulty, extreme difficulty or inability）
Cognition（MMSE） at 90±7 days after onset | at 90±7 days after onset
  Cognition is based on Mini-mental State Examination（MMSE）. （The minimum and maximum values of MMSE is 0 and 30,respectively, higher scores mean a better outcome. ）
Cognition（MoCA） at 90±7 days after onset | at 90±7 days after onset
  Cognition is based on Montreal Cognitive Assessment（MoCA）. （The minimum and maximum values of MoCA is 0 and 30,respectively, higher scores mean a better outcome.）
adverse events(AEs) and serious adverse events（SAEs) through 14 days | up to 14 days
  Any complications associated with sodium aescinate treatment (e.g. allergy, gastrointestinal complications, bleedings, thrombotic, or infectious complications) were defined as adverse events (AEs). SAEs are defined as any untoward medical occurrence or effect that at any dose results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in persistent or significant disability or incapacity. SAEs and safety endpoints are reported in line with expedited reporting regulations and then adjudicated by an independent panel.
all serious adverse events(SAEs) throughout the study follow-up period up to 3 months | up to 3 months
  SAEs are defined as any untoward medical occurrence or effect that at any dose results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in persistent or significant disability or incapacity.

CONTACTS AND LOCATIONS:
Overall Officials: Ji, Principal Investigator — Beijing Tiantan Hospital

IPD SHARING:
Plan to Share IPD: No